CLINICAL TRIAL: NCT03032185
Title: Evaluation of Effect of Transcutaneous Electrical Nerve Stimulation (TENS) on Autonomic and Psychophysical Parameters in Postmenopausal Women
Brief Title: Evaluation of the Effect of Transcutaneous Electrical Nerve Stimulation (TENS) in Postmenopausal Women
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Secretaria Municipal de Saúde de Rolante (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Lucélia Caroline dos santos Cardoso, Master of Science, Secretaria Municipal de Saúde de Rolante
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 48302915.1.0000.5307
Record Dates: First submitted 2016-01-22; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Menopause
Keywords: menopause; post-menopause; transcutaneous electrical nerve stimulation; electrical stimulation therapy; women's health
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active TENS (Active Comparator): Active TENS, 10 Hz/200 μs
  Interventions: Device: Transcutaneous Elevtrical Nerve Stimulation
- Not Active TENS (Sham Comparator): Sham TENS
  Interventions: Device: Transcutaneous Elevtrical Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Elevtrical Nerve Stimulation
  Other Names: Transcutaneous Electrical Nerve Stimulation

SUMMARY:
Introduction: Menopause is the last menstrual period, it is a natural phenomenon to all women. Postmenopausal, some women may experience unpleasant symptoms such as hot flushes, urogenital pain, headache and pains in the musculoskeletal system. That happens due to the decreased ovarian hormone secretion and changes in the autonomic system. Pain is also caused by a complex autonomic activity. For pain management, a therapeutic electrical stimulation of the peripheral nervous system promotes modulation of nociceptive incentives and release of endogenous opioids. According to reviewed studies, the use of transcutaneous electrical nerve stimulation (TENS), by directly stimulating the central nervous system, has presented results of manipulation of the autonomic system, being observed change in heart rate and cognitive improvement in dementia. Given this possibility, the present study aims to investigate whether the use of Transcutaneous Electrical Nerve Stimulation in low frequency can generate autonomic and psychophysical changes in healthy postmenopausal women.

Objective: To evaluate the effectiveness of Transcutaneous Electrical Nerve Stimulation on autonomic and psychophysical parameters in postmenopausal women.

Methods: randomized, crossover, double-blind. A sample of thirty patients will be selected according to inclusion and exclusion criteria previously established. The autonomic and psychophysical functions will be evaluated by Quantitative Sensory Testing and Conditioned Pain Modulation (pain thresholds to heat and modulation of conditioned pain, respectively), as well as scales to evaluate catastrophism and sleep quality (by scale of Pittsburgh Sleep Quality Index). After application of the scales, the participants will be subject to active Ttranscutaneous Electrical Nerve Stimulation session or sham with a fortnight washout as randomization. All the research subjects will be invited to participate in the study and sign an Informed Consent and Informed (ICI). This study will be registered in the Clinical Trials.

ELIGIBILITY:
Inclusion Criteria:

* To be in the period of post-menopause;
* Do not have chronic diseases or comorbidities in drug treatment;
* Accept to participate in the study and sign the free and informed consent form.

Exclusion Criteria:

* Start continuous medication during the study period;
* Display cognitive problems that make it difficult to understand the questionnaires and proposals;
* History of alcohol or drug abuse in the last 6 months;
* History of neurological disorders;
* History of cardiac arrhythmias;
* History of moderate or severe head injury;
* History of neurosurgery;
* Uncompensated systemic diseases, and chronic inflammatory diseases (diabetes, lupus, rheumatoid arthritis, Sjogren's syndrome, Reiter's syndrome);
* History of uncompensated hypothyroidism;
* History of personal cancer, past or treatment.
* Wish referred to leave the study at any time.
* No attendance to the stages that make up the research.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Autonomic changes in postmenopausal women's health | 30 days
  Heart rate's modification tested by R-R interval on electrocardiogram.
Psychophysical changes in postmenopausal women´s health | 30 days
  pain evaluated by Quality Sensitive Test

SECONDARY OUTCOMES:
Descendent Inibitory System Pain changes in postmenopausal women´s health | 30 days
  evaluated by conditioned pain modulated test

CONTACTS AND LOCATIONS:
Locations (1):
- Andressa de Souza, Canoas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes